CLINICAL TRIAL: NCT05910463
Title: Assessment of the Impact of the Axomove Therapy® Medical Device on Subacute or Chronic Low Back Pain Patients Leaving Rehabilitation Centres to Facilitate Self-rehabilitation: a Multicentre Randomized Controlled Study.
Brief Title: Assessing the Impact of the Axomove Therapy Medical Device on Low Back Pain Patients
Acronym: AVA-PREPA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Axomove (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KM00369
Record Dates: First submitted 2023-04-05; First posted 2023-06-18 (Actual); Last update posted 2023-07-21 (Actual); Status verified 2023-04

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AXOMOVE Therapy (Experimental): Use of a web and mobile application for remote monitoring and rehabilitation
  Interventions: Other: AXOMOVE Therapy Medical Device
- Routine care (No Intervention): Current rehabilitation support care

INTERVENTIONS:
Other: AXOMOVE Therapy Medical Device — Personalized exercise programs for the self-rehabilitation of low back pain patients
  Arms: AXOMOVE Therapy

SUMMARY:
An evaluation study of the impact of the Axomove Therapy® medical device on subacute or chronic low back pain patients leaving rehabilitation centres to facilitate self-rehabilitation. A prospective, randomized, open-label, multicentre study whose main objective is to evaluate the effectiveness of the Axomove Therapy Medical Device on disability reduction (Oswestry disability index score) patients with subacute or chronic low back pain requiring rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 18-65 years,

Patients with subacute or chronic low back pain, day hospital follow-up (HDJ) or weekday hospital with a planned return home within 2 weeks of the inclusion visit (J0), Patient with common low back pain for at least 6 weeks before hospitalization, Patient having a smartphone, tablet/ or computer (compatible with the technical requirements of the DM) and having the possibility to connect (via a telephone subscription or a WIFI connection),

Patient agreeing to install the Axomove Therapy® application and agreeing to follow the study protocol,

Patient with physical, sensory and cognitive ability to use an application (digital tools) on a smartphone, tablet or computer and perform physical exercise programs,

A patient who is a member of, or in receipt of, a social security scheme.

Exclusion Criteria:

* Patients who are unable to understand, read or speak French,

Inability to receive informed information,

A patient with a sensory, visual or tactile impairment that prevents the correct use of a smartphone, tablet and/or computer, or prevents the exercise from being carried out safely,

Patient with suspected or proven serious pathology such as recent vertebral fractures (less than 6 months), infection, malignant tumors and/or radiculopathy,

Patient with a history of rheumatic inflammatory disease,

Patient with true radiculalgia,

Patient with scoliosis > 30°, Patient with lumbar surgery in the past 12 months,

Pregnant patient, parturient or breastfeeding,

Patient under legal protection (guardianship, curatorship),

A patient with a serious and/or uncontrolled illness that, in the opinion of the investigator, could result in unacceptable safety risks or compromise protocol compliance, for example: an active or uncontrolled infection.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Estimated)
Dates: Start 2023-06-28 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Efficacy of AXOMOVE Therapy | 14 weeks (105 days)
  Functional capacity of patients measured through the Oswestry Disability Index score

SECONDARY OUTCOMES:
Level of patient physical activity | day 0 (inclusion), day 15, day 45 and day 105
  Level of physical activity measured by the international physical activity questionnaire (IPAQ-SF)
Quality of life | day 0 (inclusion), day 15, day 45 and day 105
  Quality of life measured by the EQ5D5L questionnaire
Quality of life | day 0 (inclusion), day 15, day 45 and day 105
  Quality of life measured by the SF36 questionnaire
Efficacy of AXOMOVE Therapy | day 0 (inclusion), day 15, day 45
  Functional capacity of patients measured through the Oswestry Disability Index score (ODI)

CONTACTS AND LOCATIONS:
Overall Officials: Valerie WIECZOREK, MD, Principal Investigator — CHU de Lille
Locations (1):
- CHRU de LILLE, Lille, France

IPD SHARING:
Plan to Share IPD: No